CLINICAL TRIAL: NCT00059124
Title: Aortic Calcium: Epidemiology and Progression
Brief Title: Aortic Calcium: Epidemiology and Progression -- Ancillary to MESA
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. Michael H. Criqui, Distinguished Professor, University of California, San Diego
Other Study IDs: 1213; R01HL072403 (NIH)
Record Dates: First submitted 2003-04-17; First posted 2003-04-18 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study the epidemiology of aortic calcium.

DETAILED DESCRIPTION:
BACKGROUND:

Aortic calcium measured by computed tomography occurs earlier in life than other subclinical (that is, asymptomatic) markers of cardiovascular disease (CVD), shows a wide range, and is common in women. The large size of the aorta and relative lack of image artifact from motion make it ideal for radiographic quantitative imaging. This study is ancillary to and coordinated with the Multi-Ethnic Study of Atherosclerosis (MESA), a large prospective epidemiologic study investigating multiple subclinical CVD measures and CVD risk factors. Subclinical measures in MESA include coronary calcium, carotid ultrasound, cardiac magnetic resonance imaging, and the ankle/brachial blood pressure index. The extensive CVD risk factor measurements include both traditional risk factors and newer measures such as inflammatory and genetic markers.

DESIGN NARRATIVE:

This ancillary study will determine the epidemiology of aortic calcium in 2000 randomly selected (from 6500 total) MESA participants. Questions to be addressed include predictors of aortic calcium progression; associations of aortic calcium and aortic calcium progression with other subclinical CVD measures, CVD risk factors, and demographics; and the prognostic significance of aortic calcium. The project has three primary specific aims: 1) to predict the cross-sectional aortic calcium burden as a function of other subclinical CVD measures and CVD risk factors; 2) to predict aortic calcium progression as a function of other subclinical CVD measures and CVD risk factors, and 3) to predict aortic calcium progression as a function of progression of selected subclinical CVD measures and CVD risk factors. The two secondary specific aims are 1) to contrast the results of the three primary specific aims for men vs. women, and for four major ethnic groups (White, Hispanic, Black, and Asian); and 2) to provide a database for future evaluation of whether aortic calcium and/or aortic calcium progression independently predict subsequent myocardial infarction, stroke, and other CVD events.

ELIGIBILITY:
Participation in the original MESA Study

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A random selection of approximately 1/3 of the original MESA participants.
Sampling Method: Probability Sample
Enrollment: 1980 (Actual)
Dates: Start 2003-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Abdominal Aortic Calcium | During the Exam 2 and Exam 3 MESA visits

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Criqui, MD, MPH, Principal Investigator — University of California, San Diego